CLINICAL TRIAL: NCT05224804
Title: Pharmacists' Knowledge and Attitudes About ADRs Reporting and Pharmacovigilance Practice in Egyptian Hospitals
Status: Completed | Type: Observational
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Marwa Kamal, lecturer of clinical pharmacy, phD, Fayoum University
Other Study IDs: Pharmacovigilance
Record Dates: First submitted 2022-01-29; First posted 2022-02-04 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: Adverse Drug Reaction
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: knwoledge — Knowledge and Attitudes about ADRs Reporting

SUMMARY:
The present study has assessed the knowledge, attitude and practice of ADRs reporting among pharmacists, and the perceived factors that may influence reporting.

DETAILED DESCRIPTION:
The practice and science of pharmacovigilance is described as the gathering, identification, monitoring, assessment, and prevention of adverse medication effects using pharmaceutical products. The term "pharmacovigilance" comes from the Greek words pharmakon (drug) and vigilare (vigilance) (monitor or keep an eye on). Pharmacovigilance (PV) is defined by the World Health Organization (WHO) as "the science and practices relating to the detection, assessment, understanding, and prevention of adverse effects or other drug-related problems". PV assesses the risk-benefit profile of medicines in order to improve patient safety. As a result, adverse drug reaction (ADR) reporting is the bedrock of any PV system, and early detection and reporting of ADRs to regional or national drug-regulatory bodies is important.

ADRs are defined by the World Health Organization as an unpleasant and unexpected response to a medicine that occurs at levels usually employed in man for the prevention, diagnosis, or therapy of disease, or for the alteration of physiological function". Adverse drug reactions (ADRs) are major public health issues that have been linked to longer hospital stays and higher therapeutic costs. According to recent systematic reviews and meta-analyses of observational research, the rate of hospital admissions linked to ADRs is between 3-5 percent.

A number of factors have been linked to HCPs, particularly pharmacists, reporting ADRs. Several studies have indicated reasons for not reporting observed ADRs, and pharmacists have been polled to determine the most important facilitators and barriers to spontaneous reporting. The seven deadly sins were coined by Inman and later defined by Lopez-Gonzalez et al., into professional and personal traits, as well as knowledge and attitudes toward reporting. Pharmacists from throughout the world have highlighted a number of barriers to reporting ADRs, including a lack of time, the inability to correlate an adverse event (AE) to a specific medicine, and the absence of readily available reporting forms . It has also emphasized the necessity of educational measures to encourage ADR reporting, such as awareness lectures and workshops.

Egypt joined the WHO International Program for Drug Monitoring in 2001, but no concrete actions were done until 2009, when the Egyptian Pharmacovigilance Center was established (EPVC). Receiving ADR reports, detecting safety signals, sending frequent newsletters with pharmacovigilance (PV)-related updates, and conducting awareness training are only a few of EPVC's responsibilities.

ELIGIBILITY:
Inclusion Criteria:

- Pharmacist graduates

Exclusion Criteria:

undergrauate pharmacist

-

Ages: 20 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: A total of 300 pharmacists were approached and questionnaire forms were distributed to pharmacists in different practice settings. Questionnaire was handed to them after explaining them the aim of the study. The pharmacists were asked to complete the questionnaire and hand it back after completion, Descriptive statistics including frequency and percentage was used to present the data.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-09-10 (Actual); Study Completion 2021-09-10 (Actual)

PRIMARY OUTCOMES:
Pharmacists' Knowledge and Attitudes about ADRs Reporting and Pharmacovigilance Practice in Egyptian Hospitals | 1 year and 4 month to collect data.
  The majority of pharmacists was knowledgeable about pharmacovigilance and had a favourable attitude toward ADR reporting. There are several variables that discourage pharmacists from reporting suspected ADRs, including the belief that there is no advantage to reporting, the presence of administrative barriers, the lack of availability of the ADR reporting form, and the lack of encouragement from hospital administration.

CONTACTS AND LOCATIONS:
Locations (1):
- Marwa Kamal Ahmed Tolba, Al Fayyum, Egypt

REFERENCES:
- [Background] Beninger P. Pharmacovigilance: An Overview. Clin Ther. 2018 Dec;40(12):1991-2004. doi: 10.1016/j.clinthera.2018.07.012. Epub 2018 Aug 17. PMID 30126707